CLINICAL TRIAL: NCT01640249
Title: A Single Ascending Dose, Safety, Tolerability, Pharmacokinetic, and Pharmacodynamic Study of LY3006072 in Healthy Subjects
Brief Title: A Study of LY3006072 in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated due to unacceptable pharmacokinetic (PK) profile.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 14372; I6B-MC-HZBA (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-07-11; First posted 2012-07-13 (Estimated); Results first posted 2019-08-08 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Participants received placebo capsule orally with approximately 200 to 300 milliliter (mL) of room temperature water in the morning.
  Interventions: Drug: Placebo
- LY3006072 (Experimental): Participants received LY3006072 capsules starting at 1 milligram (mg) and escalating doses of 3 mg, 10 mg, 20 mg and 40 mg.
  Interventions: Drug: LY3006072

INTERVENTIONS:
Drug: Placebo — Capsules administered orally
  Arms: Placebo
Drug: LY3006072 — Capsules administered orally
  Arms: LY3006072

SUMMARY:
The purpose of this study is to evaluate how safe LY3006072 (study drug) is and whether it causes any side effects. The study will also measure how much of the study drug gets into the blood stream and how long it takes the body to get rid of the study drug. The study drug will be given in the morning or evening with or without a meal.

This is the first time that this study drug is being given to humans. This study is for research purposes only and is not intended to treat any medical condition.

DETAILED DESCRIPTION:
This study has two parts:

Part A - single ascending dose of LY3006072 administered to healthy participants in 3 of 4 study periods (placebo in 1 of 4 periods).

Part B - morning and evening doses of LY3006072 given to healthy participants in fed and fasted states in 2 or 3 of 3 study periods (placebo in 1 of 3 periods for some participants).

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy males or females, as determined by medical history and physical examination
* Male participants with a partner of childbearing potential must agree to use barrier protection during sexual intercourse while in the study and for 3 months after the last dose of study drug
* Women must not be pregnant or nursing and must be of non-childbearing potential, due to either surgical sterilization or menopause
* Body mass index between 19.0 and 30.0 kilograms per square meter (kg/m^2), inclusive

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2012-07-24 (Actual); Primary Completion 2012-11-26 (Actual); Study Completion 2012-11-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Evansville, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a 2-part (Part A and Part B) crossover study. Part A was a dose-escalation with up to 3-period crossover with 2 alternating cohorts (Cohorts 1 and 2). There was 14 days of washout time between each dose. Part B was not initiated as study was terminated early due to technical factors.
Groups:
- Cohort 1 (Sequence 1): Participants received LY3006072 and Placebo capsules as per below dosing schedules.
  Period 1: 1 milligrams (mg) LY3006072, Period 2: 10 mg LY3006072 and Period 3: Placebo
- Cohort 1 (Sequence 2): Participants received LY3006072 and Placebo capsules as per below dosing schedules.
  Period 1: 1 mg LY3006072, Period 2: Placebo, Period 3: 40 mg LY3006072
- Cohort 1 Sequence 3: Participants received LY3006072 and Placebo capsules as per below dosing schedule.
  Period 1: Placebo, Period 2: 10 mg LY3006072 and Period 3: 40 mg LY3006072
- Cohort 1 Sequence 4: Participants received 1 mg, 10 mg and 40 mg of LY3006072 capsules as per below dosing schedule.
  Period 1: 1 mg LY3006072, Period 2: 10 mg LY3006072 and Period 3: 40 mg LY3006072
- Cohort 2 (Sequence 1): Participants received Placebo and 20 mg of LY3006072 capsules as per below dosing schedule.
  Period 1: Placebo and Period 2: 20 mg LY3006072
- Cohort 2 (Sequence 2): Participants received 3 mg and 20 mg of LY3006072 capsules as per below dosing schedule.
  Period 1: 3 mg LY3006072 and Period 2: 20 mg LY3006072
- Cohort 2 (Sequence 3): Participants received Placebo and 3 mg of LY3006072 capsules as per below dosing schedule.
  Period 1: 3 mg LY3006072 and Period 2: Placebo
Period: Period 1
Arm/Group | Cohort 1 (Sequence 1) | Cohort 1 (Sequence 2) | Cohort 1 Sequence 3 | Cohort 1 Sequence 4 | Cohort 2 (Sequence 1) | Cohort 2 (Sequence 2) | Cohort 2 (Sequence 3)
Started | 3 | 2 | 2 | 2 | 2 | 5 | 2
Received at Least 1 Dose of Study Drug | 3 | 2 | 2 | 2 | 2 | 5 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 4 | 2
Not Completed | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 1 | 0
Period: Period 2
Arm/Group | Cohort 1 (Sequence 1) | Cohort 1 (Sequence 2) | Cohort 1 Sequence 3 | Cohort 1 Sequence 4 | Cohort 2 (Sequence 1) | Cohort 2 (Sequence 2) | Cohort 2 (Sequence 3)
Started | 2 | 2 | 2 | 2 | 2 | 4 | 2
Completed | 2 | 2 | 2 | 2 | 2 | 4 | 2
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Cohort 1 (Sequence 1) | Cohort 1 (Sequence 2) | Cohort 1 Sequence 3 | Cohort 1 Sequence 4 | Cohort 2 (Sequence 1) | Cohort 2 (Sequence 2) | Cohort 2 (Sequence 3)
Started | 2 | 2 | 2 | 2 | 0 (Cohort 2 was planned for only 2 dosing periods.) | 0 (Cohort 2 was planned for only 2 dosing periods.) | 0 (Cohort 2 was planned for only 2 dosing periods.)
Completed | 2 | 2 | 2 | 1 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Cohort 1 (Sequence 3): Participants received LY3006072 and Placebo capsules as per below dosing schedule.
  Period 1: Placebo, Period 2: 10 mg LY3006072 and Period 3: 40 mg LY3006072
- Cohort 1 (Sequence 4): Participants received 1 mg, 10 mg and 40 mg of LY3006072 capsules as per below dosing schedule.
  Period 1: 1 mg LY3006072, Period 2: 10 mg LY3006072 and Period 3: 40 mg LY3006072
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (Sequence 1) | Cohort 1 (Sequence 2) | Cohort 1 (Sequence 3) | Cohort 1 (Sequence 4) | Cohort 2 (Sequence 1) | Cohort 2 (Sequence 2) | Cohort 2 (Sequence 3) | Total
Number analyzed (Participants) | 3 | 2 | 2 | 2 | 2 | 5 | 2 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 1 | 2 | 2 | 3 | 0 | 10
  >=65 years | 1 | 2 | 1 | 0 | 0 | 2 | 2 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 2 | 2 | 1 | 2 | 2 | 12
  Male | 2 | 0 | 0 | 0 | 1 | 3 | 0 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 2 | 2 | 2 | 2 | 5 | 2 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 2
  White | 2 | 2 | 2 | 2 | 2 | 4 | 2 | 16
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 2 | 2 | 2 | 2 | 5 | 2 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Drug Related Adverse Events (AEs) or Any Serious AEs
Description: AEs that were considered possibly related to study drug, in the opinion of the investigator, were reported. A summary of serious and all other non-serious AEs, regardless of possible drug relatedness, is located in the Reported Adverse Event module.
Time Frame: Baseline, up to 21 days
Population: All randomized participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo: Participants received placebo capsule orally with approximately 200 to 300 mL of room temperature water in the morning.
- 1 mg LY3006072: Participants received 1 mg LY3006072 capsule orally with approximately 200 to 300 mL of room temperature water in the morning.
- 3 mg LY3006072: Participants received 3 mg LY3006072 capsule orally with approximately 200 to 300 mL of room temperature water in the morning.
- 10 mg LY3006072: Participants received 10 mg LY3006072 capsule orally with approximately 200 to 300 mL of room temperature water in the morning.
- 20 mg LY3006072: Participants received 20 mg LY3006072 capsule orally with approximately 200 to 300 mL of room temperature water in the morning.
- 40 mg LY3006072: Participants received 40 mg LY3006072 capsule orally with approximately 200 to 300 mL of room temperature water in the morning.
Arm/Group | Placebo | 1 mg LY3006072 | 3 mg LY3006072 | 10 mg LY3006072 | 20 mg LY3006072 | 40 mg LY3006072
Number analyzed (Participants) | 9 | 6 | 6 | 6 | 6 | 6
Participants
  Serious AEs | 0 | 0 | 0 | 0 | 0 | 0
  Other Non-Serious AEs | 0 | 3 | 1 | 1 | 2 | 6

2. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY3006072
Time Frame: Predose, 0.25, 0.5, 1, 2, 3, 5, 8, 12, 16, 24, 36, 48 and 96 hours postdose
Population: All randomized participants who received at least one dose of study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | 1 mg LY3006072 | 3 mg LY3006072 | 10 mg LY3006072 | 20 mg LY3006072 | 40 mg LY3006072
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
nanograms per milliliter (ng/mL) | 18.8 (20) | 57.0 (12) | 160 (24) | 263 (42) | 576 (31)

3. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Curve (AUC) of LY3006072
Description: PK: Area Under the Concentration-Time Curve from Time Zero to Infinity (AUC[0-inf] of LY3006072.
Time Frame: Predose, 0.25, 0.5, 1, 2, 3, 5, 8, 12, 16, 24, 36, 48 and 96 hours postdose
Population: All randomized participants who received at least one dose of study drug and have evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms * hours per mL (ng*hr/mL)
Arm/Group | 1 mg LY3006072 | 3 mg LY3006072 | 10 mg LY3006072 | 20 mg LY3006072 | 40 mg LY3006072
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6
nanograms * hours per mL (ng*hr/mL) | 1530 (47) | 4800 (34) | 14400 (25) | 24700 (27) | 65600 (21)

ADVERSE EVENTS:
Time Frame: Up To 21 Days
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | Placebo | 1 mg LY3006072 | 3 mg LY3006072 | 10 mg LY3006072 | 20 mg LY3006072 | 40 mg LY3006072
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/9 | 3/6 | 1/6 | 1/6 | 2/6 | 6/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=9) | 1 mg LY3006072 (N=6) | 3 mg LY3006072 (N=6) | 10 mg LY3006072 (N=6) | 20 mg LY3006072 (N=6) | 40 mg LY3006072 (N=6)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 6 (6)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Part B was not initiated as study was terminated early due to technical factors.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days